CLINICAL TRIAL: NCT03837106
Title: Workplace Rehabilitation of Musculoskeletal Disorders in Professional Musicians: Program Optimisation and Evaluation
Brief Title: Workplace Rehabilitation for Musicians: Program Optimisation and Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Rehabilitation Department, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Musicians: RCT program #2
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation program (Experimental): Home and supervised exercise program specific to musicians. Injury prevention and management education program specific to musicians.
  Interventions: Other: Rehabilitation program
- No intervention (No Intervention): Control group, no intervention

INTERVENTIONS:
Other: Rehabilitation program — 3-month rehabilitation program comprising exercise and education specific to musicians. The program will be supported by an online platform containing more than 50 exercise videos, narrated powerpoint presentations, informative videos, quizzes, and forums for communicating with a physiotherapist and for organizing group exercise sessions.
  Arms: Rehabilitation program

SUMMARY:
Background: The classical musician's work, which comprises numerous daily hours of precise and often strenuous repetitive movements in asymmetrical postures, renders them vulnerable to musculoskeletal (MSK) injury. Performance-related MSK disorders (PRMDs) have been defined as "any pain, weakness, numbness, tingling or other physical symptoms that interfere with your ability to play your instrument at the level to which you are accustomed". The lifetime prevalence of PRMDs in professional instrumental musicians ranges from 62 to 93%. Furthermore, typical musical instruction does not include education on physical health and injury prevention, and this is thought to be an important factor in musicians' development of pain and injuries.

The combination of musician-specific exercise and education on injury prevention may have greater impacts on musicians' wellbeing than exercise or education alone. In a pilot trial, 15 orchestral musicians were offered an educational presentation and carried out a home exercise program for 11 weeks. There were no dropouts, exercise adherence was high and musicians reported improvement of their symptoms. However, certain weaknesses were identified. Thus, this type of rehabilitation program demonstrates much potential for improving the wellbeing of orchestral musicians, but improvements should be made. The collaboration of experts with relevant backgrounds, including musicians who were exposed to the program, can optimize the program.

Objectives and hypotheses: The objectives are 1) to identify facilitators and obstacles to the implementation of the initial program by realizing focus groups with musicians; 2) to adapt the program to the local context; 3) to evaluate the effectiveness of the revised program to decrease the intensity, functional impact and frequency of PRMDs in musicians with a pilot randomised controlled trial (RCT); 4) to evaluate the effect of the educational components of the program on health-related knowledge and behaviour. The hypothesis for objective 3 is that a decrease in PRMD intensity, frequency and functional limitations will be demonstrated in the experimental group following participation in the program, compared to the control group.

Methods:

1. - Focus groups: The 15 pilot project participants will be invited to share their perceptions regarding the initial program. Sessions will be comprised of questions on implementation determinants described in the Consolidated Framework for Implementation Research.
2. - Adaptation to local context: Experts in education and exercise will design the components of the program according to results from Step 1. All new or modified exercises will be reviewed by two clinicians, and tried by participants from the pilot trial. New comments will be considered, and an adapted program will be proposed.
3. - Implementation and evaluation of effectiveness Participants: Fifty orchestral musicians (25 per group) will be recruited from full and part-time orchestras and university-level music performance programs. Students will be included because the program will have the potential to directly impact the workers of tomorrow. Musicians with and without PRMDs will be invited to participate, as the program is both preventive and curative.

Study design: Pilot single-blind RCT with 1-year follow-up. Participants will be evaluated at baseline (T0), at the end of the 3-month rehabilitation program (T1) and 1 year later (T2). The baseline evaluation will consist of questionnaires on PRMD symptoms and functional limitations. Following baseline, subjects will be randomly assigned to either a rehabilitation program (exercise group) or no intervention (control group). Randomization will be stratified by instrument group and PRMD prevalence (presence or absence of symptoms). The same questionnaires will be completed by all participants at evaluations 2 and 3. All meetings will be held in participants' workplace.

Intervention: The rehabilitation program will consist of education on healthy practice habits and load and injury management and a 3-month home exercise program specific to musicians. Control group members will receive no intervention until after T2.

Baseline demographics will be compared between groups (independent t-tests, chi-square tests). Two-way mixed-model analyses of variance (ANOVA) will explore the effect of the rehabilitation program on PRMD symptoms and functional limitations.

Relevance: Orchestral musicians frequently suffer from debilitating pain that can have a lasting impact on their career. Our multi-sectorial research and clinical team hopes to create an effective rehabilitation program that can be offered to many musical populations. If the program is effective, next steps will include integration of the program into the workplace. In order to have longer-lasting and further-reaching impacts on musicians' wellbeing, the presence of rehabilitation in the workplace is the ultimate goal.

ELIGIBILITY:
Inclusion Criteria:

* Full-time classical musician with or without musculoskeletal pain, student or professional
* ≥18 years

Exclusion Criteria:

* musculoskeletal injuries non-related to musical performance
* <15 hours per week playing their instrument
* corticosteroid injection in the 6 weeks pre-recruitment
* prescribed anti-inflammatories or gabapentin in the 3 weeks pre-recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians (MPIIQM) at 12 months | Baseline, 1 year
  Self-report questionnaire containing two subscales: Pain Intensity (4 questions) and Pain Interference (5 questions). Each question is scored by the participant on a scale from 0 ("no pain" or "does not interfere" to 10 "pain as bad as you can imagine" or "completely interferes" for Pain Intensity and Pain Interference, respectively. The pain intensity scale ranges from 0 to 40, and pain interference from 0 to 50, for a possible total of 90 points (summation) where higher scores indicate worse outcomes and lower scores indicate better outcomes.

SECONDARY OUTCOMES:
Change in symptom prevalence and frequency from baseline: Nordic Musculoskeletal Questionnaire at 12 months | Baseline, 1 year
  Self-report questionnaire evaluating symptom prevalence and frequency in all regions of the body
Changes in health-related behaviour from baseline: Self-Assessment Questionnaire at 12 months | Baseline, 1 year
  Self-report questionnaire evaluating changes in health related behaviour over the course of the study
Perceived change of condition from baseline: Global Rating of Change | 1 year
  Self-report questionnaire evaluating participants' perceived change over the course of the study
Change in symptom frequency from baseline: Symptom frequency scale at 12 months | Baseline,1 year
  Self-report questionnaire evaluating frequency of symptoms on a scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- CIRRIS, Québec, Quebec, Canada

REFERENCES:
- [Derived] Roos M, Lamontagne ME, Desmeules F, Dionne C, Savard I, Pinard AM, Lafrance S, Tanguay M, Roy JS. Workplace Injury Prevention and Wellness Program for Orchestra Musicians: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2024 Sep;54(9):584-593. doi: 10.2519/jospt.2024.12277. PMID 39180194